CLINICAL TRIAL: NCT06412783
Title: Population-based Investigation of Aneurysm Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021YFC2501103
Record Dates: First submitted 2023-11-12; First posted 2024-05-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysms; Screening; Blood test
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- blood test group (Experimental)
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — performing blood tests on the participants for specific markers.

SUMMARY:
Most intracranial aneurysms are found accidentally in neurovascular imaging. And these inspection methods are limited by the problems of instrument fixation, radiation, time-consuming, contrast agent toxicity and so on. At present, blood test is an ideal alternative method for early diagnosis. Compared with imaging examination, it is economical, general screening and convenient. Blood test is simple to operate, easy to be accepted by patients, and less invasive. Early screening of aneurysms can be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-75
* Individuals with normal cognitive and communication abilities
* No serious complications, such as uncontrolled hypertension, diabetes or other chronic diseases that may affect the test results.
* Basic blood test is normal or close to normal range.

Exclusion Criteria:

* Pregnancy
* Severe heart disease, renal insufficiency, liver dysfunction and other major diseases.
* In the past 6 months, there were strokes, or other types of intracranial tumors, infections and other diseases that may affect the screening results.
* There are metal implants, including dentures, pacemakers, etc.
* Using or recently used drugs that may affect blood biomarkers ( such as anticoagulant drugs, immunosuppressive agents, etc. ).
* There are serious mental illness or cognitive dysfunction, such as claustrophobia, unable to cooperate with the completion of the test.
* It is currently participating in other clinical trials or has participated in other clinical trials in the past 3 months.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4711 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Specific markers are detected | 1hours after blood collection
  oleic acid, arachidonic acid, docasa-hexaenoic acid, interleukin 1β， interleukin 1ra, tumor necrosis factors, SOD3, PPIA, S100A8, S100A9, MPO, APOA4, THBS1.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China